CLINICAL TRIAL: NCT03914326
Title: Semaglutide Cardiovascular Outcomes Trial in Patients With Type 2 Diabetes
Brief Title: A Heart Disease Study of Semaglutide in Patients With Type 2 Diabetes
Acronym: SOUL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX9924-4473; 2018-003141-42 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1218-5368 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral semaglutide (Experimental): One tablet daily for 3.5 to 5 years
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): One tablet daily for 3.5 to 5 years
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Increasing doses (3 mg/7 mg/14 mg) of semaglutide tablets to be taken with water at the same time every morning in a fasting state
  Arms: Oral semaglutide
Drug: Placebo (semaglutide) — Placebo tablets to be taken with water at the same time every morning in a fasting state
  Arms: Placebo

SUMMARY:
The researchers are doing this study to look whether the type 2 diabetes medicine, semaglutide, has a positive effect on heart disease. Participants will either get semaglutide tablets or placebo tablets ("dummy" medicine) - which treatment is decided by chance. Participants must take one tablet with water every morning on an empty stomach and not eat or drink anything for at least 30 minutes. The study will last for about 3.5-5 years. Participants will have up to 25 clinic visits and 1 phone call with the study doctor. Women cannot be in the study if pregnant, breast-feeding or if they plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age equal to or above 50 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus
* HbA1c 6.5% - 10.0% (47 - 86 mmol/mol) (both inclusive) (latest available and no more than 30 days old local laboratory assessment based on medical records or point of care measurement)
* At least one of the below conditions (a-d):

  a) Coronary heart disease defined as at least one of the following: i. Prior myocardial infarction ii. Prior coronary revascularisation procedure iii. 50% or above stenosis in coronary artery documented by cardiac catheterisation, computerized tomography coronary angiography iv. Coronary heart disease with ischaemia documented by stress test with any imaging modality b) Cerebrovascular disease defined as at least one of the following: i. Prior stroke ii. Prior carotid artery revascularisation procedure iii.50% or above stenosis in carotid artery documented by X-ray angiography, magnetic resonance angiography, computerized tomography angiography or Doppler ultrasound c) Symptomatic peripheral artery disease (PAD) defined as at least one of the following: i. Intermittent claudication with an Ankle-brachial index (ABI) below 0.85 at rest ii. Intermittent claudication with a 50% or above stenosis in peripheral artery (excluding carotid) documented by X-ray angiography, magnetic resonance angiography, computerized tomography angiography or Doppler ultrasound iii. Prior peripheral artery (excluding carotid) revascularization procedure iv. Lower extremity amputation at or above ankle due to atherosclerotic disease (excluding e.g. trauma or osteomyelitis) d) Chronic kidney disease defined as: i. eGFR below 60 mL/min/1.73 m^2 (based on medical records using latest available and no more than 6 months old assessment)

Exclusion Criteria:

* Any of the following: myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within the past 60 days prior to the day of screening
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Heart failure presently classified as being in New York Heart Association Class IV
* Treatment with any glucagon-like peptide-1 receptor agonist within 30 days before screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9651 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (490):
- United States (91):
  - Chambliss Clinical Trials, LLC, Montgomery, Alabama
  - Medical Investigations, Inc., Little Rock, Arkansas
  - Unity Health-Searcy Medical Center, Searcy, Arkansas
  - B&K Medical Research Center, Fresno, California
  - University of Vermont Medical Center, Fullerton, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Diabetes & Endocrine Associates, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Facey Medical Foundation, Mission Hills, California
  - Monterey Endocrine & Diabetes Institute, Inc, Monterey, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - San Diego Family Care, San Diego, California
  - Lundquist Inst-Biomed Innovtn, Torrance, California
  - Coastal Metabolic Research Center, Ventura, California
  - Rocky Mount Reg VA Med-DN, Aurora, Colorado
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - New West Physicians,Inc., Golden, Colorado
  - East Coast Medical Associates, Inc., Boca Raton, Florida
  - Suncoast Clin Res Port Richey, New Port Richey, Florida
  - AdventHealth Diab Inst, Orlando, Florida
  - Ellipsis Group, Alpharetta, Georgia
  - Physicians Research Assoc. LLC, Lawrenceville, Georgia
  - Endo Res Solutions Inc, Roswell, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Rocky Mountain Diab&Osteo Ctr, Idaho Falls, Idaho
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - American Health Network of IN LLC_Franklin, Franklin, Indiana
  - American Health Network of Indiana, LLC_Greenfield, Greenfield, Indiana
  - Franciscan Health Michigan City, Michigan City, Indiana
  - American Health Network of IN LLC, Muncie, Indiana
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ileana J Tandron APMC, Slidell, Louisiana
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - Methodist Phys. Clinic, Omaha, Nebraska
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Dartmouth-Hitchcock Med Ctr, Lebanon, New Hampshire
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - AMC Community Endocrinology, Albany, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - Mountain Diabetes & Endocrine Center, Asheville, North Carolina
  - Kernodle Clin Dpt-Pvt Diagnost, Burlington, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Physicians East Endocrinology, Greenville, North Carolina
  - Eastern Nephr Assoc, PLLC, New Bern, North Carolina
  - Whiteville Medical Associates, Whiteville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Awasty Research Network,LLC, Marion, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - Twinsburg Family Health Center, Twinsburg, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Heritage Valley Medical Group Inc, Beaver, Pennsylvania
  - Primary Care Research South, Inc, McMurray, Pennsylvania
  - Aria Endocrine Metabolic Assoc, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians Inc., Pittsburgh, Pennsylvania
  - The Diabetes Center, LLC, Murrells Inlet, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Michael L Reeves, MD, Chattanooga, Tennessee
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - InvestiClin Research, Nashville, Tennessee
  - MidState Endocrine Associates, Nashville, Tennessee
  - Vanderbilt Diab Obes Clin Tri, Nashville, Tennessee
  - Trinity Clinical Research LLC, Tullahoma, Tennessee
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - Central Texas Clinical Research, Austin, Texas
  - Texas Diabetes & Endocrinology, P.A._Austin, Austin, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Synergy Groups Medical, Houston, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Midland Clinical Research Center, Midland, Texas
  - Texas Diabetes & Endocrinology, P.A._Austin, Round Rock, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Dominion Medical Associates, Richmond, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Clinical Investigation Spec. Kenosha, Kenosha, Wisconsin
- Algeria (6):
  - Internal medicine department, Algiers
  - endocrino-diabetology department, Hospital IBN BADIS., Constantine
  - Internal Medecine department CHU Ibn Badis, Constantine
  - EHU 1st November 1954, Oran
  - Internal Medicine departement CHU Oran, Oran
  - Department of internal of medicine, CHU Setif, Sétif
- Argentina (12):
  - Centro Médico CIMEL, Lanús Este, Buenos Aires
  - DIM Clinica Privada, Buenos Aires
  - Centro Medico Lebensohn, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Centro de Investigaciones Metabólicas, Capital Federal
  - Centro Diabetologico Cordoba Dr. Waitman, Córdoba
  - Centro médico privado Cemaic, Córdoba
  - Instituto Médico DAMIC, Córdoba
  - Centro Médico Privado San Vicente Diabetes, Córdoba
  - Centro Médico CIMEL, Lanús Este
  - Instituto de Investigaciones Clinicas, Mar del Plata
  - Sanatorio Britanico S.A., Rosario, Santa Fe
- Austria (5):
  - Univ.-Klinik für Innere Medizin, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Fließer-Görzer [Ordination], Saint Stefan
  - Klinik Hietzing, Vienna
  - Klinik Ottakring, Vienna
- Belgium (8):
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - UZ Antwerpen - UZA - Department of Endocrinology, Edegem
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - UZ Gent - Endocrinologie - Diabetologie, Ghent
  - AZ Groeninge - Kortrijk - Centrum Endo - Diabetologie, Kortrijk
  - UZ Leuven - Endocrinology, Leuven
  - AZ Delta - Roeselare - Diabeteskliniek, Roeselare
  - AZ Delta - Roeselare, Roeselare
- Brazil (9):
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Cline Research Center, Curitiba, Paraná
  - Quanta Diagnóstico Nuclear / Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - i9 Pesquisas Clínicas, Campinas, São Paulo
  - Instituto de Pesquisa Clinica (IPEC), São Paulo, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
- Canada (18):
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - Vancouver General Hospital_Vancouver_0, Vancouver, British Columbia
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - LMC Diabetes & Endocrinology (Barrie), Barrie, Ontario
  - LMC ClinRsrh Inc.Brampton, Brampton, Ontario
  - Aggarwal and Assoc Ltd., Brampton, Ontario
  - LMC Clinical Res Thornhill, Concord, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - My Endo Diabetes & Endo Cent, Markham, Ontario
  - Bluewater Clin Res Group, Inc., Sarnia, Ontario
  - Bluewater Clin Res Group,Inc, Sarnia, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - UHN-Toronto General Hospital, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Manna Research Mirabel, Mirabel, Quebec
  - Applied Med Inf Res, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec
- China (8):
  - Peking University People's Hospital-Endocrinology, Beijing, Beijing Municipality
  - Cangzhou People's Hospital-Endocrinology, Cangzhou, Hebei
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - The Affiliated Hospital of Jiangsu University_Zhenjiang, Zhenjiang, Jiangsu
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shanghai Fifth People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
- Colombia (6):
  - Clinica de la Costa, Barranquilla, Atlántico
  - Fundación Hospital Universidad del Norte, Soledad, Barranquilla
  - Unidad de Estudios Clínicos de la Fundación Cardiovascular de Colombia, Bucaramanga-piedecuesta, Valle Del Menzuli - Santander, Santander Department
  - Fundacion Valle del Lili, Cali, Valle del Cauca Department
  - Clinica de la Costa, Barranquilla
  - Fundación Centro de Obesidad y Metabolismo COMETA, Pasto
- Croatia (10):
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - Specijalna Bolnica Za Medicinsku Rehabilitaciju Krapinske Toplice, Krapinske Toplice
  - Klinicki bolnicki centar Osijek, Osijek
  - Opca bolnica Pula, Pula
  - KBC Rijeka, Zavod za endokrinologiju, Rijeka
  - KBC Split / Krizine / Dijabetes, Split
  - Opca bolnica Varazdin_Endocrinology, Varaždin
  - Opca bolnica Zadar_Endocrinology, Zadar
  - KB Merkur - Sveucilisna klinika Vuk Vrhovac, Zagreb
  - KB Dubrava, Zavod za endokrinologiju i dijabetes, Zagreb
- Czechia (10):
  - Fakultní nemocnice U sv. Anny v Brně, Brno
  - Intendia klinika, Chrudim
  - FN Hradec Kralove, Hradec Králové
  - Diabetologicka a Interni Ambulance MUDr. Jan Vrkoc s.r.o., Moravská Ostrava
  - Ambulance DIA - INTERNA s.r.o., Ostrava
  - Diabetologicka ambulance Plzen, Pilsen
  - MUDr. Jitka Zemanova - diabetologie a interna, s.r.o., Pilsen
  - MUDr. Jitka Zemanova diabetologie a interna, Plzeň - Východní Předměstí
  - DIALINE s.r.o., Plzeň 3
  - Institut klinicke a experimentalni mediciny_Praha, Prague
- Denmark (5):
  - Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus N
  - Bispebjerg Hospital, IC-Forskning, Copenhagen
  - Hillerød Endokrinologisk amb. H0652, Hillerød
  - Slagelse Sygehus Ambulatorium for hjertesygdomme, Slagelse
  - Svendborg Sygehus - Endokrinologisk afdeling, Svendborg
- France (8):
  - Centre Hospitalier Universitaire de Besancon-Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire de Dijon-Hopital Le Bocage, Dijon
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Assistance Publique Hopitaux de Marseille-Hopital de La Conception, Marseille
  - Centre Hospitalier de Narbonne, Narbonne
  - Ap-Hp-Hopital Bichat-Claude Bernard-1, Paris
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque-2, Pessac
  - Les Hopitaux Universitaires de Strasbourg-Hopital de Hautepierre-1, Strasbourg
- Germany (14):
  - Cardiologicum Dresden und Pirna - MVZ "Am Felsenkeller" (Dresden), Dresden
  - Uniklinik TU Dresden - Med. Klinik III, Dresden
  - Praxis Dr. med. M. Esser, Essen
  - Zentrum für klinische Forschung, Dr. med. Lüdemann, Falkensee
  - Diabetologische Schwerpunktpraxis Harburg- Dr. med.Paschen,, Hamburg
  - Diabetes Zentrum Wandsbek Berufsausuebungsgemeinschaft GbR, Hamburg
  - Praxisgemeinschaft Jerichow, Jerichow
  - Diabetologische Gemeinschaftspraxis Dr. Staudenmeyer und Dr. Schiwietz, Lingen
  - Die Praxis am Ludwigsplatz, Ludwigshafen
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
  - VvP Kliniken gGmbH Marienhospital Stuttgart - Innere Medizin I, Stuttgart
  - Forschungszentrum Ruhr KliFoCenter GmbH, Kahrmann, Witten
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- India (40):
  - Osmania General Hospital, Hyderabad, A.P.
  - Sunshine Hospital, Hyderabad, Andhra Pradesh
  - Care Outpatient Centre, Hyderabad, Andhra Pradesh
  - Ramdev Rao Hospital, Hyderabad, Andhra Pradesh
  - Apollo Excelcare Hospital, Guwahati, Guwahati, Assam
  - Apollo Excelcare Hospital, Guwahati, Assam
  - HCG Hospitals, Ahmedabad, Gujarat
  - Dr. Jivraj Mehta Health Foundation, Ahmedabad, Gujarat
  - PGIMS Rohtak, Rohtak, Haryana
  - Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - Calicut Medical College, Kozhikode, Kerala
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Goa Medical College, Goa, Maharashtra
  - P D Hinduja National Hospital and Medical Research Centre, Mumbai, Maharashtra
  - BYL Nair Hospital and T N Medical College Department of endo, Mumbai, Maharashtra
  - BSES MG hospital, Mumbai, Maharashtra
  - Fortis Hospital Mulund, Mumbai, Maharashtra
  - Fortis Hospital, Mulund, Mumbai, Mumbai, Maharashtra
  - chelleram Diabetes Institute, Pune, Maharashtra
  - Inamdar Multispeciality Hospital, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - Kanungo Institute of Diabetes Specialities Pvt Ltd, Bhubaneswar, Odisha
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Fortis Heart Institute and Multispeciality Hospital, Mohali, Punjab
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Kg Hospital and Post Graduate Medical Institute, Coimbatore, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Ranipet, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Gandhi Hospital & Medical college, Hyderabad, Telangana
  - Osmania General Hospital, Hyderabad, Telangana
  - Ramdev Rao Hospital, Hyderabad, Telangana
  - SSKM, Kolkata, West Bengal
  - Apollo Gleneagles Hospital, Kolkata, West Bengal
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - Lady Hardinge Medical College, New Delhi
  - North Delhi Diabetes Centre, New Delhi
  - Jothydev's Diabetes & Research Center, Thriruvananthapuram
- Israel (11):
  - Rambam MC - Diabetes and obesity center of excellence, Haifa
  - Hadassah Ein Karam MC - Diabetes Unit, Jerusalem
  - Clalit HMO Hamoshava Jerusalem, Jerusalem
  - Meir MC - Diabetes unit, Kfar Saba
  - Western Galilee MC - Institute of Diabetes, Nahariya
  - Rabin MC Beilinson - Endo unit, Petah Tikva
  - Sourasky MC - Institute of Endocrinology, metabolism and hypertension, Tel Aviv
  - Endrocrinolgy Clinic - Sheba Medical Center, Tel Litwinsky
  - Sheba MC - Endocrinology Clinic, Tel Litwinsky
  - Sheba MC - Cardiology Clinical Research Unit, Tel Litwinsky
  - Sheba Medica Center - Clinical Research Unit, Tel Litwinsky
- Italy (13):
  - A.O.U. Consorziale Policlinico di Bari, Bari, BA
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, Cz
  - Azienda Unita' Sanitaria Locale Toscana Nord Ovest - Cittadella della Salute Campo di Marte, Lucca, LU
  - Istituto Scientifico San Raffaele, Milan, MI
  - Policlinico Umberto I Seconda Clinica Medica, Roma, RM
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Misericordia, Perugia, Umbria
  - Università degli studi G. D'Annunzio Chieti Pescara - CAST, Chieti Scalo
  - Centro Cardiologico Monzino, Milan
  - Università Federico II Dip. di Med. Clinica e Chirurgia Ed 1, Napoli
  - Azienda Ospedaliera di Padova Malatt.Metab, Padua
  - Dip. di Medicina Interna Policlinico Universitario Palermo, Palermo
  - Policlinico Universitario Paolo Giaccone, Palermo
  - Policlinico Universitario Tor Vergata, Roma
- Japan (34):
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Jinnouchi Hospital, Kumamoto, Kumamoto, Japan
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - The University of Tokyo Hospital, Diabetes and Metabolic, Bunkyo-ku, Tokyo
  - New Tokyo Heart Clinic_Matsudo-shi, Chiba,, Chiba
  - Ehime Prefectural Central Hospital, Ehime
  - Ehime Prefectural Central Hosp, Ehime
  - Fukui Prefectural Hospital, Fukui
  - Fukuoka Tokushukai Hospital, Fukuoka
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Naka Kinen Clinic, Ibaraki
  - Uji Tokushukai Medical Center_Cardiovascular Medicine, Kyoto
  - Kyoto University Hospital, Kyoto-shi, Kyoto
  - Shinden Higashi Clinic_Miyagi, Miyagi
  - Shinshu University Hospital, Nagano
  - Saiseikai Suita Hospital, Osaka
  - Osaka University Hospital_Osaka, Osaka
  - Takatsuki Red Cross Hospital_Diabetes and Endocrine Div., Osaka
  - Takatsuki Red Cross Hospital, Osaka
  - Nozaki Tokushukai Hospital_Internal medicine, Osaka
  - Saga University Hospital, Department of Cardiology, Saga-shi, Saga
  - Hanaoka Seishu Memorial Hosp._Cardiovascular Medicine, Sapporo-shi, Hokkaido
  - Kagawa Prefectural Central Hospital, Cardiovascular Medicine, Takamatsu-shi, Kagawa
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Oyama East Clinic, Tochigi
  - Tokorozawa Heart Center, Tokorozawa-shi, Saitama
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Juntendo University Hospital_Tokyo, Tokyo
  - Juntendo University Hospital, Tokyo
  - Sugawara Clinic, Tokyo
  - Minamino Cardiovascular Hospital_Cardiovascular medicine, Tokyo
  - Minamino Cardiovascular Hospital, Tokyo
  - Tokyo Nishi Tokushukai Hospital_Cardiovascular medicine, Tokyo
  - Tokyo Nishi Tokushukai Hospital, Tokyo
- Malaysia (13):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Universiti Sains Malaysia_Kota Bharu, Kelantan, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya, Putrajaya
  - Sarawak Heart Centre, Kota Samarahan, Sarawak
  - Hospital Miri, Miri, Sarawak
  - University Technology MARA (UiTM) - Puncak Alam, Sungai Buloh, Selangor
  - University Technology MARA (UiTM) - Sg Buloh, Sungai Buloh, Selangor
  - Hospital Sultanah Bahiyah, Alor Star
  - Sarawak General Hospital, Kuching
  - Hospital Miri, Sarawak
  - Hospital Tuanku Jaafar, Seremban
- Mexico (10):
  - Inst. Jaliscience de Investigacion en Diabetes y Obesidad SC, Guadalajara, Jalisco
  - Consultorio Arechavaleta Granell María del Rosario, Guadalajara, Jalisco
  - Centro de Atención Integral al Paciente con Diabetes, Tlalpan, México, D.F.
  - Internal Medicine Clin Trials, Monterrey, Nuevo León
  - Cardiolink Clin Trials S.C., Monterrey, Nuevo León
  - Unidad Medica para la Salud Integral (UMSI), San Nicolás de los Garza, Nuevo León
  - Investigación Médica Sonora S.C., Hermosillo, Sonora
  - EME Red Hospitalaria, Mérida, Yucatán
  - Medical Care and Research S. A de C.V, Mérida, Yucatán
  - Centro de Investigación Cardiometabólica de Aguascalientes, Aguascalientes
- Netherlands (10):
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam UMC Lokatie VUMC, Amsterdam
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Reinier de Graaf Gasthuis, Delft
  - Maxima Medisch Centrum, Eindhoven
  - Martini Ziekenhuis, Groningen
  - Bethesda Diabetes Research Center en Bethesda ziekenhuis, Hoogeveen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Radboudumc, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Romania (11):
  - Clinic of Diabetes Cluj, Cluj-Napoca, Cluj
  - Spitalul Judetean de Urgenta Targoviste, Târgovişte, Dâmbovița County
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş, Mureș County
  - Sc Mediab Srl, Târgu Mureş, Mureș County
  - Novus Medical Clinica SRL, Ploieşti, Prahova
  - CMI Dr. Busegeanu Mihaela Magdalena, Ploieşti, Prahova
  - CMI Dr. Pletea Noemi SRL, Bacau
  - Diabet Med SRL, Bucharest
  - Clinical Emergency Sf. Apostol Andrei Hospital, Galati
  - Spitalul Clinic Judetean de Urgente Sf. Spiridon, Iași
  - SC Gensan SRL, Policlinica ASTRA, Sibiu
- Russia (21):
  - Tumen State Medical University, Tyumen, Russia
  - City Hospital #5, Barnaul
  - Kazan Federal University, Kazan'
  - LLC "Clinic of Aesthetic Medicine & Laser Technologies", Kazan'
  - SAHI Kuzbass Hospital(former Regional clinical hospital), Kemerovo
  - Friendship University of Russia, Moscow
  - Setchenov First Moscow State Medical University, Moscow
  - State Novosibirsk regional clinical hospital, Novosibirsk
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - SPb SBHI City Outpatient clinic #37, Saint Petersburg
  - Aurora MedFort LLC, Saint Petersburg
  - City Consultative & Diagnostic Centre #1, Saint Petersburg
  - SPb SBHI City Multifield Hospital #2, Saint Petersburg
  - Consultative & Diagnostic Center with a Outpatient Hospital, Saint Petersburg
  - Regional clinical cardiology dispensary, Saratov
  - Saratov regional clinical hospital, Saratov
  - Siberian State Medical University, Tomsk
  - Ulianovsk Regional Clinical Hospital, Ulyanovsk
  - Yaroslavl Regional Hospital, Yaroslavl
  - Polyclinic #2 in Yoshkar-Ola, Yoshkar-Ola
- Serbia (7):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocrinology department, Kragujevac
  - Clinical Centre Nis, Endocrinology, Diabetes and Metabolism, Niš
  - Policlinic for diabetes, Zaječar
- Slovakia (12):
  - Metabolicke Centrum MUDr. Katariny Raslovej s.r.o., Bratislava
  - MediTask, s.r.o, Bratislava
  - Nemocnica akademika L. Derera, UNB, Bratislava
  - HUMAN-CARE, s.r.o., Košice
  - CARDIO D&R, s.r.o., Košice
  - Nemocnica Krompachy spol. s r.o Diabetol. amb. MD Gmitrov, Krompachy
  - Diabetologicka ambulancia MUDr. Katarina Plevova, s.r.o., Nitra
  - DENTAVIA s.r.o., Poprad
  - MUDr. Jan Culak, s.r.o., Prievidza
  - Kardiologicka a interna ambulancia, Rimavská Sobota
  - Tatratrial s.r.o., Rožňava
  - IRIDIA s.r.o., Vrútky
- South Africa (14):
  - Diabetes Care Centre & CDE Centre, Benoni, Gauteng
  - Peermed Clinical Trial Centre, Johannesburg, Gauteng
  - Soweto Clinical Trial Centre, Johannesburg, Gauteng
  - Deepak Lakha, Johannesburg, Gauteng
  - Hemant Makan, Johannesburg, Gauteng
  - Centre for Diabetes, Johannesburg, Gauteng
  - Dr Seeber, Pretoria, Gauteng
  - Prof P. Joshi, Pretoria, Gauteng
  - Dr H Bacus, Berea, KwaZulu-Natal
  - Dr A Amod, Durban, KwaZulu-Natal
  - Dr T Padayachee, Durban, KwaZulu-Natal
  - Dr Pillay's Rooms, Durban, KwaZulu-Natal
  - Diabetes Clinical Trials Unit, Cape Town, Western Cape
  - UCT Clinical Research Centre, Cape Town, Western Cape
- South Korea (8):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Hanyang University GURI Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
- Spain (15):
  - Hospital Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Comarcal de Antequera, Antequera
  - Hospital del Mar, Barcelona
  - Hospital Público da Mariña, Burela de Cabo
  - Hospital Reina Sofia, Córdoba
  - Hospital Univ. de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Ribera Polusa, Lugo
  - Hospital Clinico Virgen de la Victoria, Málaga
  - Hospital Quirón, Pozuelo de Alarcón
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Virgen del Camino - Sanlúcar de Barrameda, Sanlúcar de Barrameda
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen de la Macarena, Seville
- Taiwan (3):
  - Changhua Christian Hospital_Metabolic Dept., Changhua
  - Chung Shan Medical University Hospital, Taichung
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District
- Thailand (11):
  - Songklanagarind Hospital, Songkhla, Had-Yai
  - Maharaj Nakorn Chiang Mai Hospital_Endocrilogy, Chiang Mai, Mueang Chiang Mai
  - King Chulalongkorn Memorial Hospital_Endocrinology, Bangkok
  - Police General Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital_Diabetes and Endocrinology, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital-Cardiovascular metabolic Center, Bangkok
  - SI-Dvs of Endocrinology, Bangkok
  - Siriraj Hospital-Cardio, Bangkok
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
- Turkey (Türkiye) (15):
  - T.C. Saglık Bakanlıgı Adana Sehir Egitim ve Arastirma Hastan, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Bursa Yüksek İhtisas Eğitim ve Araştırma Merkezi-Kardiyoloji, Bursa
  - T.C. Saglik Bakanligi Bursa Il Saglik Mudurlugu Yuksek Ihtıs, Bursa
  - Atatürk Üniversitesi Araştırma Hastanesi- Endokrinoloji, Erzurum
  - Eskişehir Osmangazi Üniversitesi Sağlık, Uygulama ve Araştırma Hastanesi, Eskişehir
  - Hatay Mustafa Kemal Universitesi Saglik Uygulama ve Arastirm, Hatay
  - Haseki Egitim ve Arastirma Hastanesi_ISTANBUL, Istanbul
  - Kanuni Sultan Suleyman Egitim ve Arastirma Hastanesi, Istanbul
  - Göztepe Prof. Dr.Süleyman Yalçın Şehir Hastanesi- Dahiliye, Istanbul
  - Dokuz Eylül Üniversitesi Araştırma Uygulama Hastanesi-Endokrinoloji, Izmir
  - Erciyes Üniversitesi Hastanesi- Nefroloji, Kayseri
  - Sivas Cumhuriyet Üniversitesi Hastanesi -Endokrinoloji, Sivas
  - Karadeniz University School of Medicine-Adult Endocrinology, Trabzon
  - Adana Şehir Eğitim ve Araştırma Hastanesi, Yüreğir/Adana
- Ukraine (10):
  - Cherkasy Regional Clinical Hospital - Endocrinology department, Cherkasy
  - Chernivtsi Regional Clinical Hospital - Endo Outpatient department, Chernivtsi
  - Dnipropetrovsk Regional Clinical Hospital named after І.І.Mechnikov - Endocrinology therapy department, Dnipro
  - Kyiv Railway Clinical Hospital #2 - day care department, Kyiv
  - Centre of Innovative Medical Technologies of NASU - Therapeutic and Endocrinology Department, Kyiv
  - Lviv Regional Clinical Diagnostic and Treatment Endocrinology Centre - Outpatient department, Lviv
  - Odesa Regional Clinical Hospital - Endocrinology department, Odesa
  - City Clinical Hospital #1 (Poltava) - Therapeutic department, Poltava
  - Transcarpathian Regional Clinical Hospital named after A.Novak - Endocrinology department, Uzhhorod
  - Zhytomir Regional Clinical Hospital - Endocrinology department, Zhytomyr
- United Kingdom (21):
  - Crouch Oak Family Practice, Addlestone, Surrey
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal Victoria Hospital, Belfast
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - Hathaway Surgery, Chippenham
  - WISDEM Centre, Coventry
  - Western General Hospital, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Harrogate District Hospital, Harrogate
  - Burbage Surgery, Hinckley
  - Hull Royal Infirmary, Hull
  - Royal Free - Diabetes, London
  - North Manchester General Hospital - Diabetes Centre, Manchester
  - Norfolk and Norwich University Hospital, Norfolk
  - University Dept of Medicine, Derriford Hospital, Plymouth, Plymouth
  - East Surrey Hospital, Redhill
  - The Staploe Medical Centre, Soham
  - Joint Clinical Research Facility - Swansea, Swansea

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Pop-Busui R, Rasmussen S, Deanfield JE, Buse JB, Marx N, Mulvagh SL, Inzucchi SE, Mann JFE, Emerson SS, Poulter NR, Engelmann MDM, Hovingh GK, Bayer Tanggaard K, Birkenfeld AL, Connelly KA, Haluzik M, Cavender MA, Kellerer M, Jhund PS, Gregersen S, Nielsen OW, Lam CSP, McGuire DK; SOUL Study Group. Oral Semaglutide and Heart Failure Outcomes in Persons With Type 2 Diabetes: A Secondary Analysis of the SOUL Randomized Clinical Trial. JAMA Intern Med. 2026 Feb 2:e257774. doi: 10.1001/jamainternmed.2025.7774. Online ahead of print. PMID 41627802
- [Derived] Borlaug BA, Holse C, Jung MH, Lincoff AM, Mulvagh SL, Staerk-Ostergaard J, Tuttle KR, Petrie MC. Prevalence and Associations of Systemic Inflammation in Heart Failure Across the Spectrum of Ejection Fraction. JACC Heart Fail. 2025 Oct 15:102712. doi: 10.1016/j.jchf.2025.102712. Online ahead of print. PMID 41099689
- [Derived] McGuire DK, Marx N, Mulvagh SL, Deanfield JE, Inzucchi SE, Pop-Busui R, Mann JFE, Emerson SS, Poulter NR, Engelmann MDM, Ripa MS, Hovingh GK, Brown-Frandsen K, Bain SC, Cavender MA, Gislum M, David JP, Buse JB; SOUL Study Group. Oral Semaglutide and Cardiovascular Outcomes in High-Risk Type 2 Diabetes. N Engl J Med. 2025 May 29;392(20):2001-2012. doi: 10.1056/NEJMoa2501006. Epub 2025 Mar 29. PMID 40162642
- [Derived] Marx N, Deanfield JE, Mann JFE, Arechavaleta R, Bain SC, Bajaj HS, Bayer Tanggaard K, Birkenfeld AL, Buse JB, Davicevic-Elez Z, Desouza C, Emerson SS, Engelmann MDM, Hovingh GK, Inzucchi SE, Jhund PS, Mulvagh SL, Pop-Busui R, Poulter NR, Rasmussen S, Tu ST, McGuire DK; SOUL Study Group. Oral Semaglutide and Cardiovascular Outcomes in People With Type 2 Diabetes, According to SGLT2i Use: Prespecified Analyses of the SOUL Randomized Trial. Circulation. 2025 Jun 10;151(23):1639-1650. doi: 10.1161/CIRCULATIONAHA.125.074545. Epub 2025 Mar 29. PMID 40156843
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 446 sites in 34 countries.
Pre-assignment Details: A total of 9,651 participants were enrolled/randomized (1:1) to treatment with oral semaglutide (4,825 participants) or placebo (4,826 participants). One participant was randomised twice in the trial. Thus, the FAS comprised 9,650 participants (4,825 participants in the oral semaglutide group and 4,825 participants in the placebo group).
Groups:
- Oral Semaglutide: Participants were to receive once daily semaglutide tablets with a dose escalation every 4 weeks in doses 3 mg (week 0 to week 4), 7 mg (week 4 to week 8) until maintenance dose of 14 mg was reached and maintained till the end of treatment visit (up to week 260).
- Placebo: Participants were to receive once daily placebo matching oral semaglutide until end of the treatment visit (up to week 260).
Period: Overall Study
Arm/Group | Oral Semaglutide | Placebo
Started | 4825 | 4826
Full Analysis Set | 4825 | 4825
Exposed | 4814 | 4816
Completed | 4755 | 4740
Not Completed | 70 | 86
Not completed — Withdrawal by Subject | 27 | 34
Not completed — Lost to Follow-up | 43 | 51
Not completed — Randomised more than once | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis of participants were performed on full analysis set (FAS) that was defined as all unique randomised participants and were grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide | Placebo | Total
Number analyzed (Participants) | 4825 | 4825 | 9650
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (7.6) | 66.1 (7.5) | 66.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1376 | 1414 | 2790
  Male | 3449 | 3411 | 6860
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 674 | 706 | 1380
  Not Hispanic or Latino | 4106 | 4072 | 8178
  Unknown or Not Reported | 45 | 47 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 12 | 19
  Asian | 1134 | 1121 | 2255
  Native Hawaiian or Other Pacific Islander | 4 | 5 | 9
  Black or African American | 124 | 128 | 252
  White | 3327 | 3321 | 6648
  More than one race | 185 | 192 | 377
  Unknown or Not Reported | 44 | 46 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Randomization to First Occurrence of a Major Adverse Cardiovascular Event (MACE), a Composite Endpoint Consisting of: Cardiovascular (CV) Death/Non-fatal Myocardial Infarction/Non-fatal Stroke
Description: Number of participants with first occurrence of EAC (event adjudication committee) confirmed major adverse cardiovascular event (MACE), a composite end-point. i.e., from time of randomization to first occurrence of cardiovascular (CV) death, non-fatal myocardial infarction and non-fatal stroke combined data during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 579 | 668
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Test type: Superiority — Time from randomisation to first EAC-confirmed MACE was analysed using a Cox proportional hazards model with treatment as categorical fixed factor; p = 0.0028, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.77 to 0.96]

2. Secondary Outcome: Number of Participants From Randomization to First Occurrence of CV Death;Renal Death;Onset of Persistent≥50% Reduction in eGFR(CKD-EPI);Onset of Persistent eGFR(CKD-EPI)<15 mL/Min/1.73m^2;Initiation of Chronic Renal Replacement Therapy
Description: Number of participants with first occurrence of a composite endpoint. i.e., from time of randomization to first occurrence of CV death, renal death, onset of persistent greater than or equal to (≥) 50% reduction in estimated glomerular filtration rate (eGFR) (chronic kidney disease epidemiology collaboration CKD-EPI), onset of persistent eGFR (CKD-EPI) less than (<)15 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2), initiation of chronic renal replacement therapy (dialysis or kidney transplantation) combined data during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 403 | 435

3. Secondary Outcome: Number of Participants From Randomization to Time of Occurrence of CV Death
Description: Number of participants from time of randomization to time to occurrence of EAC confirmed CV death during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 301 | 320

4. Secondary Outcome: Number of Participants From Randomization to First Occurrence of Major Adverse Limb Events (MALE), a Composite Endpoint Consisting of: Acute Limb Ischemia Hospitalisation/Chronic Limb Ischemia Hospitalisation
Description: Number of participants from randomization to first occurrence of EAC confirmed major adverse limb events (MALE), a composite endpoint consisting of: acute limb ischemia hospitalisation/chronic limb ischemia hospitalisation combined data during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 71 | 99

5. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of an Expanded MACE Composite Endpoint Consisting of: CV Death/Non-fatal Myocardial Infarction/ Non-fatal Stroke/Coronary Revascularisation/Unstable Angina Pectoris Requiring Hospitalisation
Description: The number of participants from randomisation to first occurrence of an expanded MACE composite endpoint consisting of: CV death/non-fatal myocardial infarction/ non-fatal stroke/coronary revascularisation/unstable angina pectoris requiring hospitalisation combined data during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 670 | 777

6. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of a Composite Endpoint Consisting of : All-cause Death/ Non-fatal MI/ Non-fatal Stroke
Description: The number of participants from randomisation to first occurrence of EAC confirmed composite endpoint consisting of : all-cause death/ non-fatal MI/ non-fatal stroke combined data during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 779 | 902

7. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of a Composite Heart Failure Endpoint Consisting of: CV Death/Heart Failure Requiring Hospitalisation/Urgent Heart Failure Visit
Description: Number of participants from randomisation to first occurrence of EAC confirmed composite heart failure endpoint consisting of: CV death/heart failure requiring hospitalisation/urgent heart failure visit combined data during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 405 | 443

8. Secondary Outcome: Number of Participants From Randomization to First Occurrence of CKD Endpoint:Renal Death;Onset of Persistent≥50% Reduction in eGFR (CKD-EPI);Onset of Persistent eGFR(CKD-EPI)<15 mL/Min/1.73 m^2;Initiation of Chronic Renal Replacement Therapy
Description: The number of participants from randomization to first occurrence of CKD endpoint:renal death;onset of persistent≥50% reduction in eGFR (CKD-EPI);onset of persistent eGFR(CKD-EPI)<15 mL/min/1.73 m^2;initiation of chronic renal replacement therapy combined data during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 112 | 129

9. Secondary Outcome: Number of Participants From Randomisation to Time to Occurrence of All-cause Death
Description: The number of participants from randomisation to time to occurrence of EAC confirmed all-cause death during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 528 | 577

10. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Non-fatal Myocardial Infarction (MI)
Description: The number of participants from randomisation to first occurrence of EAC confirmed non-fatal MI during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 191 | 253

11. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Non-fatal Stroke
Description: The number of participants from randomisation to first occurrence of EAC confirmed non-fatal stroke during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 144 | 161

12. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Heart Failure Requiring Hospitalisation or Urgent Heart Failure Visit
Description: The number of participants from randomisation to first occurrence of EAC confirmed heart failure requiring hospitalisation or urgent heart failure visit during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 146 | 167

13. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Coronary Revascularisation
Description: The number of participants from randomisation to first occurrence of coronary revascularisation during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 200 | 263

14. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Unstable Angina Requiring Hospitalisation
Description: The number of participants from randomisation to first occurrence of EAC confirmed unstable angina requiring hospitalisation during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 74 | 80

15. Secondary Outcome: Number of Participants From Randomisation to Time to Occurrence of Renal Death
Description: The number of participants from randomisation to time to occurrence of EAC confirmed renal death during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 1 | 7

16. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Onset of Persistent 50% or More Reduction in eGFR
Description: The number of participants from randomisation to first occurrence of onset of persistent 50% or more reduction in eGFR during in-trial period were observed. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 71 | 86

17. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Onset of Persistent eGFR (CKD-EPI) Below 15 mL/Min/1.73 m^2
Description: The number of participants from randomisation to first occurrence of onset of persistent eGFR (CKD-EPI) below 15 mL/min/1.73 m^2 during in-trial period were observed. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 23 | 33

18. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Initiation of Chronic Renal Replacement Therapy (Dialysis or Kidney Transplantation)
Description: The number of participants from randomisation to first occurrence of EAC confirmed initiation of chronic renal replacement therapy (dialysis or kidney transplantation) during in-trial period were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 40 | 48

19. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Acute Limb Ischemia
Description: The number of participants from randomisation to first occurrence of EAC confirmed acute limb ischaemia hospitalization during in-trial period were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 16 | 17

20. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of Chronic Limb Ischemia Hospitalisation
Description: The number of participants from randomisation to first occurrence of EAC confirmed chronic limb ischaemia hospitalization during in-trial period were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 63 | 88

21. Secondary Outcome: Annual Rate of Change in eGFR (CKD-EPI) (Total eGFR Slope)
Description: Annual rate of change in eGFR in terms of chronic kidney disease CKD-EPI were reported during in trial period. eGFR was calculated using the CKD-EPI formula. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 260
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization. Here 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure" also.
Measure: Mean (Standard Error); unit: ml/min/1.73 m^2 per year
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4819 | 4822
ml/min/1.73 m^2 per year | -1.67 (0.0) | -2.06 (0.0)

22. Secondary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (Week 0) up to Week 104 during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 104
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4076 | 4004
Percentage of HbA1c | -0.71 (1.22) | -0.15 (1.19)

23. Secondary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline (Week 0) up to Week 104 during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 104
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4251 | 4155
Kilograms | -4.21 (5.85) | -1.28 (4.90)

24. Secondary Outcome: Number of Severe Hypoglycaemic Episodes
Description: The number of severe hypoglycaemic episodes (such as the seriousness of hypoglycaemia, contributing factors, seizures, and unconsciousness; classified by American Diabetes Association) observed during the in-trial period were reported in this endpoint. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Episodes | 88 | 121

25. Secondary Outcome: Number of Participants From Randomisation to First Occurrence of a Severe Hypoglycaemic Episode
Description: The number of participants from randomisation to first occurrence of severe hypoglycaemic episodes (such as the seriousness of hypoglycaemia, contributing factors, seizures, and unconsciousness; classified by American Diabetes Association) during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From randomisation (week 0) up to week 265
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 4825 | 4825
Participants | 76 | 84

ADVERSE EVENTS:
Time Frame: From Week 0 up to Week 265
Description: The safety evaluation data as reported by the investigator was based on the Full Analysis Set.
Arm/Group | Oral Semaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 528/4825 | 579/4825
Serious Adverse Events (participants affected / at risk) | 2312/4825 | 2427/4825
Other Adverse Events (participants affected / at risk) | 1761/4825 | 1599/4825
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide (N=4825) | Placebo (N=4825)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 6 (7)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (2)
Abscess (Infections and infestations) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 3 (3) | 5 (5)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Abscess of external ear (Infections and infestations) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1) | 1 (1)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental death (General disorders) | 0 (0) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Acetonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 2 (2)
Acute cholecystitis necrotic (Hepatobiliary disorders) | 1 (1) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 11 (11) | 22 (24)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 123 (145) | 151 (177)
Acute left ventricular failure (Cardiac disorders) | 11 (12) | 12 (14)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 175 (196) | 229 (251)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 18 (19)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 33 (43) | 50 (61)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 11 (11)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Adenoid cystic carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (2) | 0 (0)
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 33 (39) | 44 (48)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 2 (2) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 83 (96) | 103 (111)
Angina unstable (Cardiac disorders) | 80 (97) | 104 (117)
Anginal equivalent (Cardiac disorders) | 2 (2) | 1 (1)
Angiocardiogram (Investigations) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 7 (7) | 11 (11)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Antibiotic associated colitis (Infections and infestations) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 6 (6) | 4 (5)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 0 (0) | 2 (2)
Aortic restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 2 (2)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 1 (1) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 24 (24) | 22 (22)
Aphasia (Nervous system disorders) | 2 (2) | 1 (1)
Apocrine breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Appendiceal mucocoele (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 7 (7) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 9 (9) | 7 (7)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 9 (9) | 12 (12)
Arteriosclerosis coronary artery (Cardiac disorders) | 17 (17) | 12 (12)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Arteriovenous fistula operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Arthritis bacterial (Infections and infestations) | 4 (4) | 2 (2)
Arthritis infective (Infections and infestations) | 1 (1) | 2 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 4 (5)
Aspergilloma (Infections and infestations) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 11 (11) | 10 (10)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 1 (1)
Ataxia (Nervous system disorders) | 3 (4) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atonic urinary bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrial enlargement (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 99 (106) | 95 (111)
Atrial flutter (Cardiac disorders) | 12 (14) | 11 (13)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 13 (13) | 10 (10)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 12 (12) | 6 (6)
Atypical pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 3 (3) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 13 (13)
Bacteraemia (Infections and infestations) | 6 (6) | 4 (5)
Bacterial infection (Infections and infestations) | 2 (2) | 2 (2)
Bacterial prostatitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 3 (3)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 9 (9)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0)
Basilar artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Basilar artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 1 (1) | 1 (1)
Benign biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 13 (13) | 16 (16)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 8 (8) | 6 (6)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biloma infected (Infections and infestations) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder metaplasia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (13) | 9 (9)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Bladder ulcer (Renal and urinary disorders) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister infected (Infections and infestations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 1 (1)
Blood glucose fluctuation (Investigations) | 1 (1) | 1 (2)
Blood glucose increased (Investigations) | 0 (0) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 11 (12) | 5 (5)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brachiocephalic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 9 (9) | 9 (9)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Brain injury (Nervous system disorders) | 5 (5) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 4 (4) | 6 (6)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Brainstem compression (Nervous system disorders) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 5 (7) | 10 (10)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 5 (5)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 2 (2)
Buttock injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 121 (122) | 141 (143)
COVID-19 pneumonia (Infections and infestations) | 138 (141) | 182 (186)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 2 (2)
Calculus prostatic (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 2 (2) | 2 (2)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 36 (36) | 31 (33)
Cardiac asthma (Cardiac disorders) | 2 (5) | 1 (1)
Cardiac cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 107 (141) | 116 (157)
Cardiac failure acute (Cardiac disorders) | 33 (42) | 43 (51)
Cardiac failure chronic (Cardiac disorders) | 33 (36) | 33 (38)
Cardiac failure congestive (Cardiac disorders) | 67 (78) | 58 (65)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 (0) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 20 (22) | 14 (14)
Cardiogenic shock (Cardiac disorders) | 9 (9) | 17 (17)
Cardiomegaly (Cardiac disorders) | 3 (3) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 4 (4)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 3 (3)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 2 (2)
Carotid artery disease (Nervous system disorders) | 3 (3) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 7 (7)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Carotid artery stenosis (Nervous system disorders) | 31 (31) | 19 (19)
Carpal tunnel syndrome (Nervous system disorders) | 3 (4) | 3 (3)
Cataract (Eye disorders) | 39 (46) | 49 (59)
Cataract diabetic (Eye disorders) | 1 (2) | 0 (0)
Cataract operation (Surgical and medical procedures) | 6 (6) | 2 (3)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 2 (2)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 29 (32) | 62 (71)
Cellulitis streptococcal (Infections and infestations) | 0 (0) | 2 (2)
Cement embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Cerebellar atrophy (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 3 (3) | 1 (1)
Cerebellar ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 3 (3) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral amyloid angiopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral artery occlusion (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 8 (8)
Cerebral infarction (Nervous system disorders) | 27 (28) | 30 (31)
Cerebral ischaemia (Nervous system disorders) | 7 (8) | 5 (5)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 30 (30) | 38 (40)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 4 (4) | 3 (3)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Chest pain (General disorders) | 20 (20) | 21 (21)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Cholangitis (Hepatobiliary disorders) | 6 (7) | 9 (9)
Cholangitis acute (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholangitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 17 (17) | 12 (12)
Cholecystitis acute (Hepatobiliary disorders) | 31 (36) | 19 (19)
Cholecystitis chronic (Hepatobiliary disorders) | 5 (5) | 6 (8)
Cholelithiasis (Hepatobiliary disorders) | 29 (29) | 30 (30)
Cholestasis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Chronic coronary syndrome (Cardiac disorders) | 2 (2) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 6 (6) | 3 (3)
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 31 (31) | 44 (46)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 (25) | 24 (25)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Circulatory collapse (Vascular disorders) | 3 (3) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 4 (4)
Colitis (Gastrointestinal disorders) | 9 (9) | 3 (3)
Colitis ischaemic (Gastrointestinal disorders) | 5 (5) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 4 (5) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (9)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon gangrene (Infections and infestations) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 3 (3)
Coma (Nervous system disorders) | 0 (0) | 2 (2)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 3 (3) | 1 (1)
Complication associated with device (General disorders) | 3 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (4) | 7 (7)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (10) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Coronary artery disease (Cardiac disorders) | 102 (105) | 108 (117)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 9 (10) | 11 (13)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (2) | 11 (13)
Coronary artery stenosis (Cardiac disorders) | 43 (44) | 47 (50)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Coronary vascular graft stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Craniofacial fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Craniotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Creutzfeldt-Jakob disease (Infections and infestations) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 6 (6) | 6 (6)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 2 (2)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Cystoid macular oedema (Eye disorders) | 0 (0) | 1 (1)
Cystoprostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1)
Cytotoxic lesions of corpus callosum (Nervous system disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Death (General disorders) | 43 (43) | 52 (52)
Decompression sickness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6)
Deep vein thrombosis (Vascular disorders) | 12 (12) | 11 (11)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 17 (18) | 13 (13)
Delirium (Psychiatric disorders) | 2 (2) | 7 (7)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Delusional disorder, unspecified type (Psychiatric disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 8 (9)
Dementia Alzheimer's type (Nervous system disorders) | 3 (3) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Dengue fever (Infections and infestations) | 4 (4) | 6 (6)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 1 (1)
Device loosening (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 3 (3) | 4 (4)
Device occlusion (Product Issues) | 2 (2) | 1 (1)
Device power source issue (Product Issues) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 3 (4) | 5 (6)
Device related sepsis (Infections and infestations) | 1 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 9 (9) | 16 (18)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 10 (11) | 10 (11)
Diabetic eye disease (Eye disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 20 (24) | 23 (25)
Diabetic foot infection (Infections and infestations) | 7 (8) | 8 (11)
Diabetic gangrene (Infections and infestations) | 3 (4) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 8 (8) | 13 (13)
Diabetic macroangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Diabetic nephropathy (Renal and urinary disorders) | 4 (4) | 3 (3)
Diabetic neuropathy (Nervous system disorders) | 5 (7) | 3 (3)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 1 (1)
Diabetic retinopathy (Eye disorders) | 29 (32) | 15 (16)
Diabetic vascular disorder (Vascular disorders) | 3 (3) | 2 (3)
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dialysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 10 (10)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 3 (4)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Diffuse large B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 13 (15) | 6 (7)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 14 (14) | 6 (7)
Douglas' abscess (Infections and infestations) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Dry gangrene (Vascular disorders) | 4 (4) | 6 (6)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 3 (3) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 24 (26)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Embolic cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 4 (4) | 6 (6)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Empyema (Infections and infestations) | 1 (1) | 2 (2)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 11 (11) | 8 (8)
End stage renal disease (Renal and urinary disorders) | 14 (17) | 21 (21)
Endocarditis (Infections and infestations) | 4 (4) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia with cellular atypia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 2 (3) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 7 (7) | 2 (2)
Epiglottic abscess (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 3 (5) | 2 (2)
Epiretinal membrane (Eye disorders) | 5 (5) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 5 (6) | 8 (9)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 5 (5)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 4 (4) | 6 (6)
Escherichia urinary tract infection (Infections and infestations) | 8 (8) | 7 (8)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Exercise electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Exostosis of external ear canal (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Extra-axial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Extraskeletal ossification (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 7 (7) | 3 (3)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 2 (2) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 25 (26) | 44 (50)
Fatigue (General disorders) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 10 (11) | 16 (16)
Femur fracture (Injury, poisoning and procedural complications) | 7 (7) | 23 (23)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flail chest (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Focal peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Follicular lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 2 (2)
Gallbladder abscess (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder empyema (Infections and infestations) | 4 (4) | 1 (1)
Gallbladder oedema (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 3 (3)
Gangrene (Infections and infestations) | 15 (17) | 22 (24)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 5 (5)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 5 (6) | 16 (16)
Gastritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 6 (6) | 2 (2)
Gastroenteritis (Infections and infestations) | 20 (20) | 16 (17)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 (18) | 9 (9)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 3 (3)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (2) | 2 (2)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (3) | 4 (4)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Groin abscess (Infections and infestations) | 0 (0) | 2 (2)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 1 (2)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
HER2 positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 4 (4)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 9 (9) | 8 (9)
Haemodialysis (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Haemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 10 (10) | 6 (6)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 6 (7) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 14 (14) | 6 (6)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Heart failure with midrange ejection fraction (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure with preserved ejection fraction (Cardiac disorders) | 4 (4) | 4 (4)
Heart failure with reduced ejection fraction (Cardiac disorders) | 6 (6) | 7 (7)
Heart valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Heart valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hemiataxia (Nervous system disorders) | 0 (0) | 1 (1)
Hemihyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 3 (3)
Hemiplegia (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 8 (8) | 6 (6)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 3 (3)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic infarction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 2 (3) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 2 (2)
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (14) | 12 (12)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herpes sepsis (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 10 (10) | 14 (15)
Hodgkin's disease nodular sclerosis stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 6 (6) | 16 (16)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 7 (7)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 38 (45) | 41 (49)
Hyperglycaemic crisis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 5 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (12) | 32 (37)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 13 (13) | 20 (22)
Hypertensive crisis (Vascular disorders) | 12 (13) | 6 (6)
Hypertensive emergency (Vascular disorders) | 3 (6) | 6 (6)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hypertensive end-organ damage (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 2 (2) | 0 (0)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 9 (12) | 5 (5)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 10 (15) | 8 (12)
Hypnic headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 37 (45) | 44 (51)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 2 (2) | 2 (2)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 12 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (9) | 12 (12)
Hypoosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 27 (27) | 9 (9)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Hypothyroidic goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 5 (5) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
IVth nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 6 (7) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 3 (3) | 4 (5)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 3 (3) | 0 (0)
Impaired healing (General disorders) | 4 (4) | 2 (2)
Implant site dehiscence (General disorders) | 0 (0) | 1 (1)
Implantable defibrillator replacement (Surgical and medical procedures) | 2 (2) | 0 (0)
Incarcerated hernia (General disorders) | 2 (2) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 2 (2) | 2 (2)
Infection (Infections and infestations) | 3 (3) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 10 (10) | 7 (7)
Inguinal hernia (Gastrointestinal disorders) | 28 (29) | 15 (16)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 7 (9) | 4 (6)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 18 (20) | 7 (7)
Intervertebral discitis (Infections and infestations) | 3 (3) | 2 (2)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal angina (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 5 (6)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 (7) | 14 (14)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 8 (8) | 7 (7)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 3 (3)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (1)
Ischaemic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 65 (72) | 59 (67)
Jaundice (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 0 (0) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Kidney congestion (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 3 (3) | 4 (4)
Knee arthroplasty (Surgical and medical procedures) | 3 (3) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Lacunar infarction (Nervous system disorders) | 2 (2) | 7 (7)
Lacunar stroke (Nervous system disorders) | 3 (3) | 4 (4)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 6 (6) | 10 (12)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 0 (0) | 3 (3)
Left ventricular dysfunction (Cardiac disorders) | 3 (3) | 2 (2)
Left ventricular failure (Cardiac disorders) | 3 (3) | 6 (6)
Leg amputation (Surgical and medical procedures) | 1 (1) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lens disorder (Eye disorders) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukoplakia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 3 (3) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 5 (5) | 5 (5)
Loss of consciousness (Nervous system disorders) | 3 (4) | 3 (3)
Loss of personal independence in daily activities (Social circumstances) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 6 (6) | 5 (5)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (14)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (5)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 7 (7)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1)
Macular hole (Eye disorders) | 2 (2) | 1 (1)
Macular oedema (Eye disorders) | 3 (4) | 2 (2)
Magnesium metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 4 (4) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Malignant ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (6)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 3 (3) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Medical device site inflammation (General disorders) | 1 (1) | 0 (0)
Medical device site joint pain (General disorders) | 0 (0) | 1 (1)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 4 (4)
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Meningitis leptospiral (Infections and infestations) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Mental status changes (Psychiatric disorders) | 11 (14) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 9 (9) | 11 (11)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 6 (6) | 10 (11)
Metabolic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Metapneumovirus pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 9 (9)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1) | 3 (3)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 5 (5)
Mitral valve repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Mixed dementia (Nervous system disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Morganella infection (Infections and infestations) | 0 (0) | 1 (1)
Motor neurone disease (Nervous system disorders) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 14 (14) | 11 (11)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Mycobacterium chelonae infection (Infections and infestations) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelopathy (Nervous system disorders) | 1 (1) | 4 (4)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial bridging (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 3 (3) | 3 (3)
Myocardial infarction (Cardiac disorders) | 40 (40) | 47 (48)
Myocardial ischaemia (Cardiac disorders) | 25 (26) | 46 (52)
Myocardial rupture (Cardiac disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Myopericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Narcolepsy (Nervous system disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 20 (21) | 13 (14)
Nephropathy (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Neurosurgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Non-Hodgkin's lymphoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 39 (43) | 24 (25)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Normochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 5 (5) | 5 (5)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ocular myasthenia (Eye disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 3 (3)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 5 (5) | 4 (4)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 10 (10) | 6 (6)
Osteitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 39 (41) | 58 (66)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Osteomyelitis (Infections and infestations) | 12 (13) | 22 (26)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 4 (4)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 2 (3) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 3 (3) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Otolithiasis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Pacemaker syndrome (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Palpitations (Cardiac disorders) | 0 (0) | 5 (5)
Pancreatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pancreatic cyst (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Pancreatic neuroendocrine tumour metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 16 (16) | 14 (18)
Pancreatitis chronic (Gastrointestinal disorders) | 4 (4) | 5 (6)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Paracancerous pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 4 (4)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 2 (2)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Parietal lobe stroke (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 4 (4)
Paronychia (Infections and infestations) | 3 (3) | 1 (1)
Parotid abscess (Infections and infestations) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 3 (3) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Pelvic mass (General disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 1 (1) | 0 (0)
Penile vascular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (4) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 5 (5)
Perihepatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 60 (72) | 64 (75)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 15 (16) | 11 (12)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 11 (13) | 11 (13)
Peripheral artery thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Peripheral circulatory failure (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 21 (23) | 17 (21)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral nerve lesion (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 6 (6) | 8 (9)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritoneocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 7 (7)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Peyronie's disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 2 (2) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 15 (16)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 129 (146) | 129 (148)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 11 (11) | 15 (15)
Pneumonia bacterial (Infections and infestations) | 19 (23) | 12 (13)
Pneumonia chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia legionella (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 2 (3) | 0 (0)
Pneumonia viral (Infections and infestations) | 8 (8) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Polyp (General disorders) | 0 (0) | 1 (1)
Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Porcelain gallbladder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 3 (3) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 2 (2) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 8 (9) | 7 (7)
Presyncope (Nervous system disorders) | 5 (5) | 4 (4)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Procedural shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 40 (40) | 23 (23)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 7 (7)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Prostatic abscess (Infections and infestations) | 1 (1) | 4 (4)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 6 (6) | 3 (3)
Prostatomegaly (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Prosthetic cardiac valve malfunction (Product Issues) | 1 (1) | 0 (0)
Prosthetic cardiac valve regurgitation (General disorders) | 1 (1) | 0 (0)
Prosthetic cardiac valve stenosis (General disorders) | 0 (0) | 2 (2)
Prosthetic valve endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pseudohyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 1 (2) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 19 (20)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 18 (20)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 2 (5) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 0 (0)
Purulent discharge (Infections and infestations) | 0 (0) | 1 (1)
Pyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 7 (7) | 10 (13)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 6 (6)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 1 (1) | 1 (1)
Pyomyositis (Infections and infestations) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 15 (15) | 6 (6)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 8 (8) | 5 (6)
Rectal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 2 (2)
Renal artery stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal atrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Renal colic (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 9 (10) | 9 (10)
Renal impairment (Renal and urinary disorders) | 11 (11) | 7 (7)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 27 (28)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 1 (1)
Retinal detachment (Eye disorders) | 4 (4) | 2 (2)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 2 (2) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Retinopathy proliferative (Eye disorders) | 0 (0) | 3 (5)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Revascularisation procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 12 (12) | 14 (14)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 12 (12) | 10 (10)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (10)
Rotator cuff tear arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SARS-CoV-2 sepsis (Infections and infestations) | 0 (0) | 3 (3)
Sacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 1 (1)
Scalp haematoma (Vascular disorders) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 7 (7) | 4 (6)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scrotal cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Scrub typhus (Infections and infestations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 7 (10) | 8 (9)
Senile dementia (Nervous system disorders) | 2 (2) | 2 (2)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 50 (57) | 43 (46)
Septic arthritis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 22 (22) | 32 (32)
Serratia infection (Infections and infestations) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 3 (3) | 3 (3)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 3 (3)
Shoulder fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 5 (5)
Sinus node dysfunction (Cardiac disorders) | 7 (7) | 8 (8)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 12 (13) | 17 (20)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleeve gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 6 (7)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 2 (2) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Spigelian hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (4)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 2 (2)
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (7)
Spinocerebellar disorder (Nervous system disorders) | 1 (1) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1)
Splenic artery perforation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spondylectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 6 (6)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 5 (5) | 3 (3)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Starvation ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Stent malfunction (Product Issues) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Streptococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Streptococcal sepsis (Infections and infestations) | 3 (3) | 2 (2)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 6 (7) | 7 (7)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 4 (4)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 12 (14) | 9 (9)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Subgaleal haematoma (Vascular disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 9 (9) | 10 (10)
Sudden death (General disorders) | 17 (17) | 19 (19)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 2 (2)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Supraventricular bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 6 (6) | 4 (4)
Suspected COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 37 (42) | 35 (36)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 5 (5) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 5 (5) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Third degree chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 2 (2) | 3 (3)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Thymic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 2 (2) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Tobacco abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Tolosa-Hunt syndrome (Eye disorders) | 2 (2) | 0 (0)
Tongue carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 3 (3)
Tractional retinal detachment (Eye disorders) | 1 (1) | 1 (1)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 42 (51) | 43 (48)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 4 (4)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Trifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 2 (3) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 3 (4) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tumefactive multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 (4) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 (7) | 3 (3)
Ulcer (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 7 (7)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 5 (5)
Upper limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 9 (10)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 4 (4) | 4 (4)
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urethrotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 11 (11) | 9 (11)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 63 (69) | 62 (70)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 17 (18) | 23 (25)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
VIth nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 2 (2) | 2 (5)
Varicophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 2 (2) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular calcification (Vascular disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 4 (4) | 2 (2)
Vascular device infection (Infections and infestations) | 2 (2) | 2 (3)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vascular graft infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Vascular graft restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular stenosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 2 (3) | 3 (3)
Vascular stent stenosis (General disorders) | 7 (8) | 9 (9)
Vascular stent thrombosis (General disorders) | 5 (6) | 0 (0)
Vasodilation procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 4 (4) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 6 (6) | 5 (5)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 9 (9)
Ventricular septal defect acquired (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 13 (16) | 20 (21)
Vertebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 1 (2)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar stroke (Nervous system disorders) | 1 (1) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 9 (9) | 9 (9)
Vertigo positional (Ear and labyrinth disorders) | 4 (4) | 4 (4)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 2 (2) | 3 (3)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 11 (11) | 9 (10)
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (16) | 7 (7)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Wound cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 5 (5) | 5 (5)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide (N=4825) | Placebo (N=4825)
COVID-19 (Infections and infestations) | 756 (838) | 777 (836)
Diabetic retinopathy (Eye disorders) | 943 (1122) | 932 (1116)
Nausea (Gastrointestinal disorders) | 344 (442) | 62 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT03914326/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03914326/SAP_001.pdf